CLINICAL TRIAL: NCT02147938
Title: French Multicentre Observational Study of a Prospective Cohort of Renal Transplant Patients Converted From the Twice Per Day Form of Tacrolimus (Prograf®) to the Once Per Day Form (Advagraf®)
Brief Title: A Study of Renal Transplant Patients Converted From the Twice Per Day Form of Tacrolimus (Prograf®) to the Once Per Day Form (Advagraf®)
Acronym: OPALE
Status: Completed | Type: Observational
Sponsor: Astellas Pharma S.A.S. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: FR-ADV-NI-003
Record Dates: First submitted 2014-05-15; First posted 2014-05-28 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Renal Transplantation
Keywords: France; Tacrolimus; Prograf; Observational; Advagraf
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: early conversion from Prograf® to Advagraf®: patients converted during the first 6 months post-transplantation
  Interventions: Drug: Tacrolimus
- 2: late conversion from Prograf® to Advagraf®: patients converted between 6 and 12 months post-transplantation
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Advagraf®; Prograf®; FK506

SUMMARY:
Assessment in a real situation of the conversion conditions, the efficacy and the safety of the treatment with tacrolimus in renal transplant patients converted from the tacrolimus twice per day form (Prograf®) to the tacrolimus once per day form (Advagraf®) with follow-up at one year.

Analysis of two groups of patients: patients converted from Prograf® to Advagraf® early (during the first 6 months post-transplantation) or late (between 6 and 12 months post-transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patient for less than one year
* Patient where the conversion from Prograf® to Advagraf® has been decided by the doctor

Exclusion Criteria:

* Patient participating in an interventional clinical trial at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Tacrolimus daily dose conversion ratio (mg Prograf® / mg Advagraf®) | At baseline (i.e. time of conversion)
  Percentage of patients with a tacrolimus dose conversion ratio of 1mg / 1mg and percentage of patients with a ratio ≠ 1mg / 1mg
Time to measurement of the first trough tacrolimus blood concentration (C0) after conversion | From baseline (conversion) to first determination of C0 assessed up to one year
  number of days between the date of conversion and the date of first assay of C0 after conversion
Number of additional visits that the doctor considers to be due to the conversion (if applicable) | At 6 months and at 1 year follow-up visit
  percentage of patients with additional visit(s) and percentage of patients without additional visit

SECONDARY OUTCOMES:
Reasons for the conversion | At baseline
  number of capsules, poor treatment compliance, requested by patient, safety, centre practice, other
Profile of the patients in both groups | At baseline
  sociodemographic data, transplantation history, comorbidities, post-transplantation complications, risk factors and concomitant treatments (Immunosuppressive protocols (IS) and others) at the time of conversion and changes, if applicable, at 6 months and 1 year post-conversion
Time to reach steady state | Time from baseline (conversion) to steady state C0 assessed up to one year
Dose ratio at steady state | At baseline (conversion) and up to 6 months post-baseline
  calculation of the tacrolimus daily dose ratio once the steady state is reached: mg Prograf® at conversion / mg Advagraf® once the steady state is reached. Percentage of patients with a ratio of 1mg / 1mg and percentage of patients with a ratio ≠ 1mg / 1mg.
The intra-patient variability (IPV) of tacrolimus | At baseline and up to 6 months post-baseline
Latest available laboratory data with Prograf® before conversion and with Advagraf® | At baseline, 6 months and 1 year follow-up visit
  Values and dates for blood and urine renal parameters, blood glucose
Compliance with the treatment at conversion and at 1 year post-conversion | At baseline and 1 year follow-up visit
  Compliance with the treatment at conversion (taking Prograf®) and at 1 year post-conversion (taking Advagraf®) only in group 2 (late conversion) will be assessed using the Morisky questionnaire, from which a score will be calculated
The quality of life of the patient at conversion and at 1 year post-conversion | At baseline and 1 year follow-up visit
  The quality of life of the patient at conversion (taking Prograf®) and at 1 year post-conversion (taking Advagraf®) only in group 2 (late conversion) will be assessed using the EQ5D-5L questionnaire
Incidence of biopsy proven acute rejections (BPAR) and survival of the graft and of the patient | At 1 year follow-up visit
Occurrence of adverse effects | From baseline until 1 year follow-up visit after baseline (conversion)

CONTACTS AND LOCATIONS:
Overall Officials: Medical and Scientific Affairs Manager, Transplantation, Study Director — Astellas Pharma S.A.S.
Locations (26):
- France (26):
  - Site, Amiens
  - Site, Angers
  - Site, Besançon
  - Site, Brest
  - Site, Caen
  - Site, Clermond-Ferrand
  - Site, Créteil
  - Site, Dijon
  - Site, Le Krémlin-Bicêtre
  - Site, Lille
  - Site, Limoges
  - Site, Lyon
  - Site, Marseille
  - Site, Montpellier
  - Site, Nancy
  - Site, Nantes
  - Site, Nice
  - Site, Paris
  - Site, Poitiers
  - Site, Rennes
  - Site, Rouen
  - Site, Saint-Etienne
  - Site, Strasbourg
  - Site, Suresnes
  - Site, Toulouse
  - Site, Tours

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.